CLINICAL TRIAL: NCT06449079
Title: Predictive Risk Algorithm for Development of Right Ventricular Pacing Induced Cardiomyopathy - a Step Towards Personalized Pacemaker Lead Deployment
Brief Title: The PICM Risk Prediction Study - Application of AI to Pacing
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 333705
Record Dates: First submitted 2024-03-25; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure; Pacemaker-Induced Cardiomyopathy; Pacemaker Complication
MeSH Terms: conditions — Heart Failure | interventions — Machine Learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pacing induced cardiomyopathy: Patients who received a pacing device and developed pacing induced cardiomyopathy
  Interventions: Other: Machine learning
- Non-pacing induced cardiomyopathy: Patients who received a pacing device and did not develop pacing induced cardiomyopathy
  Interventions: Other: Machine learning

INTERVENTIONS:
Other: Machine learning — Analysis of data with machine learning methods

SUMMARY:
Development of pacing induced cardiomyopathy (PICM) is correlated to a high morbidity as signified by an increase in heart failure admissions and mortality. At present a lack of data leads to a failure to identify patients who are at risk of PICM and would benefit from pre-selection to physiological pacing. In the light of the foregoing, there is an urgent need for novel non-invasive detection techniques which would aid risk stratification, offer a better understanding of the prevalence and incidence of PICM in individuals with pacing devices and the contribution of additional risk factors.

DETAILED DESCRIPTION:
Retrospective review of patient characteristics including 12 lead resting electrocardiograms and imaging data (CMR, CT, echo, CXR and fluoroscopy of pacing leads) of patients with right sided ventricular pacing lead due to symptomatic bradycardia, who developed pacing induced cardiomyopathy (or need for CRT upgrade) versus patients who did not using supervised machine learning methods. Development of personalised predictive pacing algorithm to improve right ventricular lead placement, such as conduction system pacing or pre-emptive implantation of an additional left ventricular lead to prevent left ventricular dilatation and pacemaker-induced cardiomyopathy (PICM) with heart failure (left ventricular ejection fraction <50% by Simpson method), hospitalisation or death with the use of the retrospective patient data through machine learning.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received a pacing device (VVI, DDD, ICD, leadless pacemaker) from the GSTT/RBH/KCH/ICH database in the last 10 years (from 01/01/2014)
* All patients who are >18 years old.
* Male and Female

Exclusion Criteria:

* Patients who did not receive a pacing device (VVI, DDD, ICD, leadless pacemaker)
* All patients <18 years old
* Patients with congenital heart disease
* Patients who have received artificial heart valves or underwent cardiac bypass surgery
* Patients who did not have an echocardiogram after receiving a pacing device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who received a pacemaker at GSTT and RBH in the last 10 years and all patients who received a pacemaker at KCH and ICH in the last 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary aim | 2.5 years
  Number of risk factors in participants who developed pacing induced cardiomyopathy

SECONDARY OUTCOMES:
Secondary aim | 2.5 years
  1. To establish, through the GSTT/RBH/KCH/ICH RV-paced study population the prevalence of pacemaker induced cardiomyopathy (PICM)
Tertiary aim | 2.5 years
  2. To establish, through the GSTT/RBH/KCH/ICH RV-paced study population the incidence of PCIM 2. To establish, through the GSTT/RBH/KCH/ICH RV-paced study population the incidence of PCIM
Quarternary aim | 2.5 years
  3.• To establish mortality of PICM
Quinary aim | 2.5 years
  4. To establish the morbidity of PICM
Senary aims | 2.5 years
  5.• To include predictive value for pacing induced cardiomyopathy risk with combination of imaging data of right ventricular lead position or leadless pacemaker position
Septenary aim | 2.5 years
  6.• To include predictive value for pacing induced cardiomyopathy risk with combination of imaging data of myocardial pathology from echocardiogram and cardiac MRI

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Guys' and St Thomas' Hospital NHS Trust, London
  - Kings' College London Healthcare Trust, London
  - Imperial College London Healthcare Trust, London

IPD SHARING:
Plan to Share IPD: No